CLINICAL TRIAL: NCT05581797
Title: Psilocybin-assisted Interpersonal Therapy for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Otago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UOtagoPsilocybin
Record Dates: First submitted 2022-10-02; First posted 2022-10-17 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-04

CONDITIONS: Depressive Disorder, Treatment-Resistant
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Psilocybin-assisted psychotherapy (Experimental): Interpersonal Therapy integrated with psilocybin
  Interventions: Other: Psilocybin-assisted psychotherapy

INTERVENTIONS:
Other: Psilocybin-assisted psychotherapy — 8 sessions of interpersonal therapy and 2 doses of psilocybin

SUMMARY:
This is a single-arm, open-label interventional study of psilocybin-assisted interpersonal therapy for treatment resistant depression. 20 participants will be recruited to take part in this 8-week intervention that involves 8 sessions of psychotherapy and 2 doses of psilocybin.

DETAILED DESCRIPTION:
Study Design Interventional, Single arm, open label

1. Hypotheses:

1. It is feasible to deliver Psilocybin treatment integrated into interpersonal therapy for people with treatment resistant major depression (TRD).
2. It is feasible to recruit patients with TRD for this treatment in New Zealand.

2. Participants The study will recruit 20 participants who have a current diagnosis of Treatment resistant Major Depressive Disorder. The participants will need to agree to cease psychotropic medications including antidepressants as part of the preparation for psilocybin dosing.

3. Recruitment Participants will be recruited by referral from mental health services, primary care and community advertisements.

4. Screening

Screening involves a two-step process:

1. Participants will register their interest via a secure online Redcap website that will ask questions regarding initial eligibility. Those who pass the initial online screening and consent to further assessment of eligibility will be screened via telephone and review of online health records to determine whether they meet major inclusion/exclusion criteria, and thus whether they are eligible for an in-person screening session.
2. In-person screening will include a history and physical examination, ECG, a 30 cc blood draw for study measures and medical screening, a personal and family medical history questionnaire, psychiatric /psychological assessments and urine drug and pregnancy tests. These will be performed by clinical staff in the Clinical Research Unit (CRU, University of Otago, Christchurch Whatu Ora Waitaha).

5. Clinical assessment Psychiatric screening will be conducted by structured assessments Structured Clinical Interview for DSM Disorders (SCID), (mood and substance use sections) by the study team. After this screening potential participants will be clinically assessed by a consultant psychiatrist on the team, who will oversee participants care throughout the study and will liaise with the participants current health provider regarding the study, antidepressant discontinuation, clinical progress and any support required at the conclusion of the study. Psychoactive drug-use history, history of antidepressant treatments, and information about employment status and current functioning (including mood and psychological and psychosomatic symptoms) will be obtained.

Participants will be required to refrain from illicit drug use during the course of the study, and a urine test will be conducted before each psilocybin dosing session (e.g., testing for various opioids, stimulants and sedatives). Pregnant or nursing women are ineligible; female participants will receive a urine pregnancy test at intake and before each drug session and must agree to use effective methods of contraception during the study.

6. Informed consent process Written informed consent will be obtained at the Clinical Research Unit at the start of the in-person screening.

7. Intervention The study intervention is described in detail in the Interpersonal Therapy (IPT)+ Psilocybin Manual and is modified from Yale Manual for Psilocybin-assisted Therapy of Depression and Protocol for 'Effects of Psilocybin therapy for major depressive disorder: randomized clinical trial'. The intervention involves 8 sessions of psychotherapy and two doses of psilocybin over 10 weeks and one follow-up session at 18 weeks in the Clinical Research Unit, Dept of Psychological Medicine, University of Otago, Christchurch. During the study period (week 0-9) the participants will be under the care of the consultant psychiatrists and clinical team at the Clinical Research Unit, this includes the planned weekly contact as well as provision of urgent care during hours (via a duty clinician and psychiatrist), and the Crisis Resolution Team (CDHB) after hours.

Following screening and baseline measurements antidepressants will be gradually discontinued and Interpersonal Therapy (IPT) will be commenced in preparation for psilocybin dosing. Antidepressant discontinuation will follow clinical guidelines and will be supervised by consultant psychiatrist on the team, who will oversee participants care throughout the study. The discontinuation schedule is initial dropping of dose by half followed by tapering over 2-6 weeks. The 3 IPT preparation sessions are designed around the beginning phase of IPT (timeline of stressors and mood episodes, interpersonal inventory and identification of psychotherapy focus). The next sessions will involve psilocybin dosing and debriefing (2 psilocybin dosing sessions and 1 debriefing). This will be followed by 5 integration sessions of IPT. The IPT integration sessions will formulate the psilocybin experience within an IPT framework. IPT utilises emotional processing to facilitate change and it is anticipated this will be intensified in the psilocybin sessions.

Consultant psychiatrists will review each participant after completing psychotherapy to assess participants' ongoing treatment needs, including recommencing antidepressant medication if needed and referral to specialist mental health service if required.

ELIGIBILITY:
1. Able to give written informed consent
2. Have a confirmed DSM-5 diagnosis of Major Depressive Disorder and currently experiencing a major depressive episode and no improvement despite two adequate courses of antidepressant treatment of different pharmacological classes lasting at least 6 weeks within the current depressive episode
3. Have a baseline total score of >13 on HAMD17 .
4. Agree to discontinue any recommended psychoactive medications, including antidepressants and lithium as part of the study.
5. Agree to refrain from using alcohol and other substances including nicotine, within 24 hours of each drug administration.
6. Be judged by study team clinicians to be at low risk for suicidality
7. Be medically stable as determined by screening for medical problems via a personal interview, a medical questionnaire, a physical examination, an electrocardiogram (ECG), and routine medical blood and urinalysis laboratory tests
8. Agree to consume approximately the same amount of caffeine-containing beverage (e.g., coffee, tea) that he/she consumes on a usual morning, before arriving at the research unit on the mornings of drug session days.
9. Agree not to take sildenafil (Viagra®), tadalafil, or similar medications within 72 hours of each drug administration.
10. Agree that for one week before each drug session, he/she will refrain from taking any non-prescription medication, nutritional supplement, or herbal supplement except when approved by the study investigators. Exceptions will be evaluated by the study investigators and will include acetaminophen, non-steroidal anti-inflammatory drugs, and common doses of vitamins and minerals.
11. If female, they must agree to pregnancy testing and regular contraception while in study.
12. Have limited lifetime use of hallucinogens (the following criteria are preferred: no use in the past 5 years; total hallucinogen use less than 10 times)
13. Agree to participate in a 10-week combined psychotherapy and psilocybin intervention, complete required measurements (including follow-up measures at week 18) and adhere to safety protocols.

Exclusion Criteria:

1. Women who are pregnant (as indicated by a positive urine pregnancy test assessed at intake and before each drug session) or nursing; women who are of child-bearing potential and sexually active who are not practicing an effective means of birth control.
2. Cardiovascular conditions: coronary artery disease, stroke, angina, uncontrolled hypertension, a clinically significant ECG abnormality (e.g., atrial fibrillation), prolonged QTc interval (i.e., QTc > 450 msec), artificial heart valve, or TIA in the past year
3. Epilepsy with history of seizures
4. Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of hypoglycemia
5. Currently taking psychoactive prescription medication on a regular (e.g., daily) basis which are unable to be ceased (under supervision) during the study period.
6. Currently taking on a regular (e.g., daily) basis any medications having a primary centrally-acting serotonergic effect, including MAOIs. For individuals who have intermittent or PRN use of such medications, psilocybin sessions will not be conducted until at least 5 half-lives of the agent have elapsed after the last dose.
7. Current or past history of meeting DSM-5 criteria for schizophrenia spectrum or other psychotic disorders (except substance/medication-induced or due to another medical condition), or Bipolar I or II Disorder
8. Current or history within one year of meeting DSM-5 criteria for a moderate or severe alcohol or other drug use disorder (excluding caffeine)
9. Have a first or second-degree relative with schizophrenia spectrum or other psychotic disorders (except substance/medication-induced or due to another medical condition), or Bipolar I or II Disorder
10. Has a psychiatric condition judged to be incompatible with establishment of rapport or safe exposure to psilocybin
11. History of a medically significant suicide attempt
12. Has failed to respond to electroconvulsive therapy during the current major depressive episode 13Not fluent in English

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
The feasibility of delivery of Psilocybin integrated into Interpersonal Therapy for people with TRD | Week 10
  Retention rate (participants who complete the full number of treatment sessions).
The feasibility of recruiting patients with major depression for this treatment in New Zealand | Week 0
  1. The percentage of potential participants who meet the major inclusion/exclusion criteria during phone screening.
  2. The percentage of potential participants who enter the study after the in-person screening (see page 2 for description of two-step screening process).

SECONDARY OUTCOMES:
GRID-Hamilton Depression Rating Scale (GRID-HAMD) | Completed at baseline, week 1,2,3,4,5,6,7,8,9,18
  This scale assesses severity of depressive symptoms with a higher score indicating more severe depression. Min 0 Max 68
Social Adjustment Scale - Modified (SAS-M) | This will be completed at baseline, prior to first dosing, weeks 9 and 18.
  Measures selected interpersonal functioning items from the social adjustment scale with higher scores indicating lower interpersonal functioning. Min 24 Max 120
Therapy Goals Measurement (TGM) | This will be completed at week 2, 9 and 18.
  Measures goals participants may wish to achieve from participating in therapy. Min 4 Max 40. Higher scores indicate higher goal acheivement.
Antidepressant Discontinuation Symptom Measurement (ADSM) | This will be completed at week 1,2, and 3.
  Assesses the seven most common symptoms associated with antidepressant medication discontinuation. Min 5 Max 35. Higher scores indicate more severe withdrawal symptoms
Aotearoa Adapted Watts Connectedness Scale (AA-WCS). | At the end of psilocybin dosing session in Week 4 and Week 5
  Measures sense of connectedness to self, others, and world. HIgher scores indicate higher degrees of connectedness
Revised Mystical Experiences Questionnaire (MEQ30) | At the end of psilocybin dosing session in Week 4 and Week 5
  A measure of mystical experiences during psilocybin. Min 0 Max 150. Higher scores indicate greater intensity of mystical experiences
Qualitative interview | Week 18
  Participants' views on the number of treatment sessions, timing of psilocybin dosing. This will be used to determine if changes to the number and timetable of sessions are required

CONTACTS AND LOCATIONS:
Overall Officials: Cameron Lacey, PhD, Principal Investigator — University of Otago
Locations (1):
- University of Otago, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davis AK, Barrett FS, May DG, Cosimano MP, Sepeda ND, Johnson MW, Finan PH, Griffiths RR. Effects of Psilocybin-Assisted Therapy on Major Depressive Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2021 May 1;78(5):481-489. doi: 10.1001/jamapsychiatry.2020.3285. PMID 33146667